CLINICAL TRIAL: NCT00924612
Title: Phase II Study of the Effect of Food With Various Levels of Fat on the Pharmacokinetics of an Oral Testosterone Undecanoate Formulation in Hypogonadal Men
Brief Title: Study to Determine the Effect of Food on the Absorption of an Oral Testosterone Undecanoate Formulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLAR-09008
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Male Hypogonadism
Keywords: Primary hypogonadism; Secondary hypogonadism
MeSH Terms: conditions — Eunuchism; Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: Open-label, five-period, randomized, four-sequence (ABCDE, BDCEA,CBEDA, DBAEC), cross-over study to determine the effect of food containing various amounts of dietary fat on the pharmacokinetics of oral TU.
Oversight: Data Monitoring Committee: No

ARMS (5):
- Fasting (Treatment A) (Experimental): Single dose of oral testosterone undecanoate (containing 300 mg T) administered orally in a fasted state
  Interventions: Drug: Oral testosterone undecanoate (containing 300 mg T)
- Very low fat diet (Treatment B) (Experimental): Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with very low fat (6-10% fat).
  Interventions: Drug: Oral testosterone undecanoate (containing 300 mg T)
- Low fat diet (Treatment C) (Experimental): Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with low fat (20% fat).
  Interventions: Drug: Oral testosterone undecanoate (containing 300 mg T)
- Normal diet (Treatment D) (Experimental): Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with normal fat (30% fat).
  Interventions: Drug: Oral testosterone undecanoate (containing 300 mg T)
- High fat diet (Treatment E) (Experimental): Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with high fat (50% fat).
  Interventions: Drug: Oral testosterone undecanoate (containing 300 mg T)

INTERVENTIONS:
Drug: Oral testosterone undecanoate (containing 300 mg T)

SUMMARY:
The purpose of the study is to determine the effect of food with various amounts of fat on the absorption of an oral testosterone undecanoate formulation.

DETAILED DESCRIPTION:
Pharmacokinetics will be evaluated after the following types of meals: very low fat, low fat, normal diet, high fat, and fasting. Subjects will have one dose of TU administered 30 minutes after the initiation of the meal.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-65
* Morning serum testosterone (T) <300 ng/dL on two occasions

Exclusion Criteria:

* Significant intercurrent disease
* Abnormal prostate digital rectal exam, elevated PSA, AUA symptom score >15 or history of prostate cancer.
* Serum transaminases >2 times upper limit of normal
* Serum bilirubin >2.0 mg/dL
* Hematocrit <35% or >50%
* BMI >36
* Untreated, obstructive sleep apnea.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Swerdloff, MD, Principal Investigator — LABiomedical Research Institute at Harbor-UCLA Medical Center
Locations (2):
- LABiomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California, United States
- Anapharm, Inc., Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen subjects (8 at each study center) were enrolled. A total of 72 subjects were screened (16 subjects at the Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center and 56 subjects were screened at Anapharm, beginning on April 3, 2009.
Groups:
- Sequence ABCDE: Fasting (Treatment A) followed by dose-associated breakfast meals comprised of ~ 800 calories consisting of very low fat (6-10% fat; Treatment B), low fat (20% fat; Treatment C), "normal diet" (30% fat; Treatment D), and high fat (50% fat; Treatment E).
  Participants received a single dose of oral testosterone undecanoate (containing 300 mg T) administered in the fasted state and at 30 minutes after the initiation of protocol-defined breakfasts. Treatments were separated by 7 days.
- Sequence BDCEA: Dose-associated breakfast meals comprised of ~ 800 calories consisting of very low fat (6-10% fat; Treatment B), followed by "normal diet" (30% fat; Treatment D), low fat (20% fat; Treatment C), high fat (50% fat; Treatment E) and fasting (Treatment A).
  Participants received a single dose of oral testosterone undecanoate (containing 300 mg T) administered in the fasted state and at 30 minutes after the initiation of protocol-defined breakfasts. Treatments were separated by 7 days.
- Sequence CBEDA: Dose-associated breakfast meals comprised of ~ 800 calories consisting of low fat (20% fat; Treatment C), followed by very low fat (6-10% fat; Treatment B), high fat (50% fat; Treatment E) "normal diet" (30% fat; Treatment D), and fasting (Treatment A).
  Participants received a single dose of oral testosterone undecanoate (containing 300 mg T) administered in the fasted state and at 30 minutes after the initiation of protocol-defined breakfasts. Treatments were separated by 7 days.
- Sequence DBAEC: Dose-associated breakfast meals comprised of ~ 800 calories consisting of "normal diet" (30% fat; Treatment D), followed by very low fat (6-10% fat; Treatment B), fasting (Treatment A), high fat (50% fat; Treatment E) and low fat (20% fat; Treatment C), Participants received a single dose of oral testosterone undecanoate (containing 300 mg T) administered in the fasted state and at 30 minutes after the initiation of protocol-defined breakfasts. Treatments were separated by 7 days.
Period: Overall Study
Arm/Group | Sequence ABCDE | Sequence BDCEA | Sequence CBEDA | Sequence DBAEC
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross over design in which each enrolled subject participated in each arm in a randomized order.
Groups:
- All Study Participants: Single dose of oral testosterone undecanoate (containing 300 mg T) administered orally in a fasted state (Treatment A) and followed by a dose-associated breakfast meal comprised of ~800 calories consisting of very low fat (6-10% fat, Treatment B), low fat (20% fat, Treatment C), normal diet (30% fat, Treatment D) and high fat (50% fat, Treatment E). Participants were randomized to one of the 4 treatment sequences (ABCDE, BDCEA, CBEDA, OR DBAEC).
  Oral testosterone undecanoate (containing 300 mg T)
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 8
  United States | 8
Height [Mean (Standard Deviation); unit: centimeters] | 174.1 (7.7)
Weight [Mean (Standard Deviation); unit: kilograms] | 91.1 (14.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Mean T Cavg25 Following Meals Containing Various Amounts of Dietary Fat Compared to Normal Fat Diet
Description: PK population where subjects are randomly assigned to one of four dietary sequences of five fat regimens. Active drug is identical for all subjects and all diets. Effect of normal dietary fat is compared to fasting, very low fat, low fat, and high fat diets for mean T Cavg25.
Time Frame: 25 hour serial blood draws separated by 4 to 10 days of washout between treatments.
Population: PK population
Measure: Geometric Mean (Standard Deviation); unit: ng/dL
Groups:
- Fasting: Single dose of oral testosterone undecanoate (containing 300 mg T) administered orally in a fasted state
  Oral testosterone undecanoate (containing 300 mg T)
- Very Low Fat Diet: Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with very low fat (6-10% fat).
  Oral testosterone undecanoate (containing 300 mg T)
- Low Fat Diet: Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with low fat (20% fat).
  Oral testosterone undecanoate (containing 300 mg T)
- Normal Diet: Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with normal fat (30% fat).
  Oral testosterone undecanoate (containing 300 mg T)
- High Fat Diet: Single dose of oral testosterone undecanoate (containing 300 mg T) administered, 30 minutes after the initiation of protocol-defined breakfast of ~800 calories with high fat (50% fat).
  Oral testosterone undecanoate (containing 300 mg T)
Arm/Group | Fasting | Very Low Fat Diet | Low Fat Diet | Normal Diet | High Fat Diet
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
ng/dL | 6.38 (0.456) | 6.73 (0.410) | 6.88 (0.356) | 7.00 (0.264) | 7.18 (0.312)
Statistical Analysis 1: Comparison: Normal Diet vs High Fat Diet; Comparison of diets based on full crossover model; Test type: Other; p = 0.0025, t-test, 2 sided; Odds Ratio, log = 130.83, 90% CI 2-sided [113.59 to 150.70], Standard Error of Mean 0.0844; ANOVA of a multicenter, 4 sequence, 5 treatment crossover model using ln-transformed data. Normal fat diet compared to fasting, very low fat, low fat, and high fat diets as part of the overall analysis. No adjustments for multiplicity made
Statistical Analysis 2: Comparison: Low Fat Diet vs Normal Diet; Comparison of diets based on full crossover model; Test type: Other; p = 0.8494, t-test, 2 sided; Odds Ratio, log = 101.84, 90% CI 2-sided [86.80 to 119.47], Standard Error of Mean 0.0954
Statistical Analysis 3: Comparison: Very Low Fat Diet vs Normal Diet; Comparison of diets based on full crossover model; Test type: Other; p = 0.0013, t-test, 2 sided; Odds Ratio, log = 73.55, 90% CI 2-sided [63.23 to 85.55], Standard Error of Mean 0.0902
Statistical Analysis 4: Comparison: Fasting vs Normal Diet; Comparison of diets based on full crossover model; Test type: Other; p < 0.0001, t-test, 2 sided; Odds Ratio, log = 62.62, 90% CI 2-sided [53.38 to 76.46], Standard Error of Mean 0.0954

ADVERSE EVENTS:
Time Frame: 3 months
Description: Throughout the study, subjects were monitored for AEs. At the beginning of each study period, after the subject had had an opportunity to spontaneously mention any problems, the Principal Investigator, or nominee, inquired about AEs by asking standard questions.
Arm/Group | Fasting | Very Low Fat Diet | Low Fat Diet | Normal Diet | High Fat Diet
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 0/16 | 2/16 | 4/16 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasting (N=16) | Very Low Fat Diet (N=16) | Low Fat Diet (N=16) | Normal Diet (N=16) | High Fat Diet (N=16)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otopharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes